CLINICAL TRIAL: NCT01325064
Title: Central and Peripheral Blood Pressure and Its Relation With Vascular Target Organ Damage in Carotid, Retinal and Arterial Stiffness. Developed and Validation of a Tool
Brief Title: Blood Pressure and Subclinical Organ Damage
Acronym: Vasorisk
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: GRS 498/A/10
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: Carotid Artery Diseases; Blood Pressure; Blood Pressure Monitoring, Ambulatory; Peripheral Vascular Diseases; Retinal Vessels
MeSH Terms: conditions — Diabetes Mellitus; Carotid Artery Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: The purpose of this study is to analyze the relationship between central and peripheral blood pressure (clinic and ambulatory) with vascular structure and function, assessed by carotid intima-media thickness (IMT), artery venous retinal index, pulse wave velocity (PWV) and ankle-brachial index in patients with diabetes type 2 and without diabetes type 2. Develop and validate a software to measure the retinal vessels and to estimate arterio-venous index automatically.

Methods/design: The investigators will Perform a coss-sectional study with control group, with follow-up of 4 years in primary care. The study population will be diabetic type 2 patients with a control group without diabetes mellitus. The investigators will include by consecutive sampling 300 patients between 34 and 75 and without previous cardiovascular disease, half of each group. Main measurements: age, sex, height, weight and waist circumference. Lipids, creatinine, microalbuminuria, blood glucose, HbA1C, insulin, fibrinogen, hs-CRP and markers of endothelial dysfunction. Clinic and ambulatory blood pressure (MAPA). Ultrasonography to assess carotid IMT, retinography to assess arterio-venous ratio. ECG to evaluate left ventricular hypertrophy, ankle-brachial index and morphology analysis (PWA) and pulse wave velocity (PWV) in Sphigmocor System.

Discussion: The investigators provide information regarding various parameters derived from MAPA and pulse wave analysis of with target organ damage, especially with the vascular structure and function assessed by IMT and PWV and endothelial dysfunction in patients with diabetes type 2 and without this disease. The investigators also hope to demonstrate the usefulness of the tool developed for automatic evaluation of retinal vascularization in the early detection of abnormalities of vascular structure and function and the prognosis of cardiovascular disease in the medium term.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 34 years or more but less than 75 years, with and without type 2 diabetes.

Exclusion criteria:

* Patients who fail to meet the requirements of the protocol (mental disorders and / or cognitive uncooperative, education and understanding limitations),
* Patients with ischemic heart disease, cerebrovascular disease or other atherosclerotic disease
* Patients who are participating or will participate in a clinical trial during the study
* Patients with serious comorbidity that might endanger his life in the next 12 months.

Ages: 34 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be diabetic type 2 patients with a control group without diabetes mellitus. We will include by consecutive sampling 300 patients between 34 and 75 and without previous cardiovascular disease, half of each group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
subclinical organ damage | december, 1 2013

CONTACTS AND LOCATIONS:
Overall Officials: Manuel A Gomez, Study Director — Infoslaud Fundation
Locations (1):
- Luis Garcia Ortiz, Salamanca, Spain

REFERENCES:
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Fernandez-Alonso C, Martinez Vizcaino V, Cantera CM, Guenaga-Saenz N, Gonzalez-Viejo N, Garcia-Ortiz L; EVIDENT Study, Spain. Electrocardiographic left ventricular hypertrophy criteria and ambulatory blood pressure monitoring parameters in adults. Am J Hypertens. 2014 Mar;27(3):355-62. doi: 10.1093/ajh/hpt198. Epub 2013 Nov 4. PMID 24190901
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Gomez-Sanchez L, Gomez-Sanchez M, Garcia-Ortiz L; Vasorisk group. Relationship between uric acid and vascular structure and function in hypertensive patients and sex-related differences. Am J Hypertens. 2013 May;26(5):599-607. doi: 10.1093/ajh/hps097. Epub 2013 Feb 26. PMID 23443729
- [Derived] Garcia-Garcia A, Garcia-Ortiz L, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Gomez-Marcos MA. Relationship of 24-h blood pressure variability with vascular structure and function in hypertensive patients. Blood Press Monit. 2013 Apr;18(2):101-6. doi: 10.1097/MBP.0b013e32835ebc58. PMID 23388405
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Rodriguez-Sanchez E, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Martin C, Castano-Sanchez C, Runkle I, Gomez-Marcos MA. Sodium and potassium intake present a J-shaped relationship with arterial stiffness and carotid intima-media thickness. Atherosclerosis. 2012 Dec;225(2):497-503. doi: 10.1016/j.atherosclerosis.2012.09.038. Epub 2012 Oct 5. PMID 23084712
- [Derived] Garcia-Garcia A, Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Rodriguez-Sanchez E, Agudo-Conde C, Garcia-Ortiz L; Vaso-risk group. Office and 24-hour heart rate and target organ damage in hypertensive patients. BMC Cardiovasc Disord. 2012 Mar 22;12:19. doi: 10.1186/1471-2261-12-19. PMID 22439900
- [Derived] Recio-Rodriguez JI, Gomez-Marcos MA, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Garcia-Ortiz L; Vaso-Risk group. Cocoa intake and arterial stiffness in subjects with cardiovascular risk factors. Nutr J. 2012 Feb 10;11:8. doi: 10.1186/1475-2891-11-8. PMID 22325068
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Parra-Sanchez J, Gonzalez Elena LJ, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Gomez-Marcos MA; Vaso-risk group. A new tool to assess retinal vessel caliber. Reliability and validity of measures and their relationship with cardiovascular risk. J Hypertens. 2012 Apr;30(4):770-7. doi: 10.1097/HJH.0b013e3283506628. PMID 22306849
- [Derived] Recio-Rodriguez JI, Gomez-Marcos MA, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Garcia-Ortiz L; Vasorisk group. Abdominal obesity vs general obesity for identifying arterial stiffness, subclinical atherosclerosis and wave reflection in healthy, diabetics and hypertensive. BMC Cardiovasc Disord. 2012 Feb 1;12:3. doi: 10.1186/1471-2261-12-3. PMID 22292502
- [Derived] Garcia-Ortiz L, Ramos-Delgado E, Recio-Rodriguez JI, Agudo-Conde C, Martinez-Salgado C, Patino-Alonso MC, Rodriguez-Sanchez E, Gomez-Marcos MA; Vaso risk group. Peripheral and central arterial pressure and its relationship to vascular target organ damage in carotid artery, retina and arterial stiffness. Development and validation of a tool. The Vaso risk study. BMC Public Health. 2011 Apr 27;11:266. doi: 10.1186/1471-2458-11-266. PMID 21524299